CLINICAL TRIAL: NCT00981825
Title: Efficacy of Salivary Bacteria and Post Brushing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ER0-2007-SAL-01-GX
Record Dates: First submitted 2008-09-26; First posted 2009-09-22 (Estimated); Results first posted 2009-09-22 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Salivary Bacteria Levels
MeSH Terms: interventions — Fluorides; Triclosan; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): fluoride toothpaste control
  Interventions: Drug: Fluoride
- B (Active Comparator): triclosan/fluoride toothpaste
  Interventions: Drug: Triclosan/Fluoride

INTERVENTIONS:
Drug: Fluoride — Whole mouth brushing for 7 days
  Other Names: fluoride toothpaste (Colgate Great Regular Flavor toothpaste)
  Arms: A
Drug: Triclosan/Fluoride — Brush whole mouth twice daily for 7 days
  Other Names: triclosan/fluoride toothpaste (Colgate Total toothpaste)
  Arms: B

SUMMARY:
Research study to compare the effects of brushing with two commercially available toothpastes on salivary bacteria after brushing

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers 18-65 years of age
* Good general health
* Must sign informed consent form
* Must discontinue oral hygiene on the mornings of each appointment and between sampling periods.
* No history of allergy to personal care consumer products, or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study.

Exclusion Criteria:

* Medical condition which requires pre-medication prior to dental procedures/visits
* Medical condition which precludes eating/drinking for 12 hrs.
* History of allergy to common dentifrice ingredients
* Subjects unable or unwilling to sign the informed consent form.
* Moderate or advanced periodontal disease.
* 2 or more decayed untreated dental sites at screening.
* Other disease of the hard or soft oral tissues.
* Impaired salivary function (e.g. Sjogren's syndrome or head and neck irradiation).
* Use of medications that can currently affect salivary flow
* Current use of antibiotics
* Use of antibiotics or antimicrobial drugs within 30 days prior to study visit #1.
* Pregnant or nursing women.
* Participation in any other clinical study within 30 days prior to enrollment into this study.
* Use of tobacco products
* Subjects who must receive dental treatment during the study dates.
* Current use of Antibiotics for any purpose.
* Immune compromised individuals (HIV,AIDS, immuno suppressive drug therapy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neelim Utgikar, DDS, Principal Investigator
Locations (1):
- India GTC, Colgate Palmolive(I) ltd, Mumbai, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At clinical site
Groups:
- Fluoride 1st , Triclosan/Fluoride 2nd: Fluoride toothpaste (placebo)used in first period, then washout of 7 days, then Triclosan/Fluoride in second period.
- Triclosan/Fluoride 1st, Fluoride 2nd: Triclosan/Fluoride toothpaste (experimental)used in first period,washout of 7 days, then Fluoride in second period.
Period: First Intervention
Arm/Group | Fluoride 1st , Triclosan/Fluoride 2nd | Triclosan/Fluoride 1st, Fluoride 2nd
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Washout After 1st Intervention
Arm/Group | Fluoride 1st , Triclosan/Fluoride 2nd | Triclosan/Fluoride 1st, Fluoride 2nd
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Fluoride 1st , Triclosan/Fluoride 2nd | Triclosan/Fluoride 1st, Fluoride 2nd
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fluoride 1st, Triclosan/Fluoride 2nd: Fluoride toothpaste (placebo)
- Triclosan/Fluoride 1st, Fluoride 2nd: Triclosan/Fluoride toothpaste (experimental)
- Total: Total of all reporting groups
Arm/Group | Fluoride 1st, Triclosan/Fluoride 2nd | Triclosan/Fluoride 1st, Fluoride 2nd | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.8 (6.8) | 30.5 (8.7) | 30.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  India | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: CFU (Colony Forming Units)
Description: Total number of salivary bacterial colony forming units (lower number = less colonies present)
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: number of colony forming units
Groups:
- Fluoride Toothpaste (Control): Fluoride toothpaste (control)
- Triclosan/Fluoride Toothpaste: Triclosan/Fluoride toothpaste (experimental)
Arm/Group | Fluoride Toothpaste (Control) | Triclosan/Fluoride Toothpaste
Number analyzed (Participants) | 22 | 22
number of colony forming units | 7.18 (0.61) | 6.94 (0.40)
Statistical Analysis 1: Comparison: Fluoride Toothpaste (Control) vs Triclosan/Fluoride Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 16 days
Arm/Group | Fluoride 1st , Triclosan/Fluoride 2nd | Triclosan/Fluoride 1st, Fluoride 2nd
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days